CLINICAL TRIAL: NCT02084602
Title: Assessment of in Vivo and in Vitro Efficacy of Combined Artesunate/Mefloquine Therapy for Treatment of Uncomplicated Plasmodium Falciparum Infection in the Peruvian Amazon
Brief Title: Assessment of Artesunate/Mefloquine in the Peruvian Amazon
Acronym: Artesunate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Salud. Peru (Other Government)
Collaborators: U.S. Naval Medical Research Unit No.6 (NAMRU-6) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U.2012.0008
Record Dates: First submitted 2014-03-07; First posted 2014-03-12 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Malaria, Falciparum
Keywords: artesunate; mefloquine; falciparum; peruvian amazon
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artesunate; Mefloquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Artesunate/mefloquine (Experimental): Orally administration of artesunate 4mg/Kg by three days Orally administration of mefloquine 15mg/Kg in the fourth day Orally administration of mefloquine 10mg/Kg in the fifth day
  Interventions: Drug: Artesunate; Drug: Mefloquine

INTERVENTIONS:
Drug: Artesunate — Orally administration of artesunate 4mg/Kg by three days
  Other Names: Distribuited by AC Farma
Drug: Mefloquine — Orally administration of mefloquine 15mg/Kg in the fourth day Orally administration of mefloquine 10mg/Kg in the fifth day
  Other Names: Distribuited by AC Farma

SUMMARY:
There is growing evidence of the emergence of P. falciparum resistance to artesunate (a derivative of artemisin) in Southeast Asia. The emergence and spread of resistant strains to artemisinin would represent an alarming threat to the success of the antimalarial combination therapy in the region. The delayed clearance of parasitemia for more than 24 hours has been taken as an early sign of resistance, a phenomenon seen at the Thai-Cambodia border.

The purpose of this research study, is to assess the in vitro and in vivo efficacy of combinated artesunate/mefloquine therapy to treatment of uncomplicated Plasmodium falciparum malaria in the Peruvian Amazon through the analysis of the rate of clearance of parasitemia and other important outcomes.

DETAILED DESCRIPTION:
Combination therapy with artemisinin derivatives is the treatment of choice for malaria by P. falciparum since 2006, but there is growing evidence of the emergence of P. falciparum resistance to artesunate in Southeast Asia. The delayed clearance of parasitemia for more than 24 hours has been taken as an early sign of resistance, a phenomenon seen at the Thai-Cambodia border. The emergence and spread of resistant strains to artemisinin would represent an alarming threat to the success of the antimalarial combination therapy in the region.

This research study, will be conducted in collaboration with the National Institute of Health of Peru.

Objectives:

Main Objective: To determine the rate of clearance of parasitemia in the first 72 hours after administration of artesunate.

Secondary/exploratory objectives:

1. to determine the efficacy of the artesunate (AS)/mefloquine (MQ) therapy in participants with uncomplicated falciparum malaria in the Peruvian Amazon (sub-study);
2. to correlate the clinical results from the in vivo study with results of in vitro sensitivity and molecular genotyping;
3. to identify common specific genetic determinants to the resistance of artemisinins in parasite populations;
4. to determine the levels of gametocytes in participants with uncomplicated falciparum malaria treated with AS/MQ;
5. to determine the contribution of host immunity in clinical and parasitological response;
6. to create a catalog of parasite samples closely correlated with clinical response data to perform a longitudinal follow-up of resistance trends;
7. to determine pharmacokinetic parameters associated with failure of therapy.

Methodology:

The study will be conducted in seven health facilities and one hospital in the Department of Loreto in the Peruvian Amazon, where 59 volunteers will be enrolled between 5 and 65 years of age with confirmed diagnosis of monoinfection by P. falciparum. In addition to the main study, we will conduct a sub-study to determine the efficacy of AS/MQ (regime currently used in Peru) After signing the informed consent/assent, blood samples will be taken to determine parasite density, baseline biochemical tests, genotyping studies, analysis of molecular markers and in vitro sensitivity, antibodies against malaria and cytokines. Artesunate will be administered according to national guidelines in the first three days, 4 mg/kg/day. However, mefloquine administration will be delayed for up to 72 hours to measure the rate of clearance of parasitemia with artesunate alone in the first three days. Serial blood samples for thick/thin smears will be taken every 4 hours during the first 12 hours and then every 6 hours until complete the first 72 hours, after the AS administration, during which time the study participants will remain in a hospital ward. Monitoring will be undertaken until day 42 with analysis of thick/thin smears according to WHO guidelines. In case of parasitemia recurrence, additional blood samples will be collected for genotyping tests, in vitro sensitivity, and analysis of molecular markers of drug resistance and immunology assays. The sub-study will be useful to assess the efficacy of the regimen currently in use by the Ministry of Health of Peru, in this arm the patients will be given AS 4 mg/kg/day in Days 0, 1 and 2 and MQ 12.5mg/kg/day in Days 1 and 2. In this arm, the follow up will be done using thick smears on Days 1, 2, 3, 7, 14, 21, 28, 35 and 42. Blood samples will be collected on Days 0, 42 and the day of recurrence.

This study will allow the Ministry of Health to know the state of resistance/tolerance to artesunate in Peru and take the necessary control measures to ensure that artesunate can be used successfully for treatment of falciparum malaria. Importantly, the results of this study will be compared to parallelly-designed studies in Kenya (US Army Medical Research Unit Kenya-USAMRU K) and Thailand (Army Forces Medical Research Institute of Medical Sciences-AFRIMS).

Relevance: Malaria is one of the main public health problems in Peru, early and efficacious treatment in the principal control strategy the appearance of strains that are resistant to the regular treatment used in Peru jeopardize the strategies for malaria control in South America. This study will allow us to know the current resistance status and to prepare corresponding measures.

Budget: This study will be done as a joined effort between NAMRU-6 and the INS, this will cost 201,934.93 Nuevos Soles afforded by Instituto Nacional de Salud and a total cost of 527,934.93 Nuevos Soles for both participating institutions

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 65 years old inclusive
* Monoinfection of P. falciparum confirmed by microscopy
* Documented fever (axillary temperature > 37.5°C) and/or history of fever during the previous 48 hours in the absence of other obvious causes of fever (such as pneumonia, otitis media, etc)
* Infection with P. falciparum of 1000 and 100,000 asexual parasites per microliter (μl) to be determined by microscopic examination of a thick or thin smear, and positive confirmation by polymerase chain reaction (PCR); * Presence of sexual form of P. vivax is acceptable; ** PCR confirmation is not an enrollment requirement
* Informed consent must be obtained from the participant or both parents/guardian (in the case of children), and assent from the child (from 8 to 17 years old)
* Willingness of the participant to return to the health facility for regular check-ups during the follow-up period of 42 days
* Willingness of the participant to transfer to the Hospital de Apoyo Iquitos to start treatment

Exclusion Criteria:

* Severe malaria signs (as defined by the World Health Organization):

  1. Cerebral malaria (irreversible coma)
  2. Severe anemia (hematocrit < 15%, or clinic signs)
  3. Clinic signs of kidney failure (e.g., serum creatinine > 3 mg/dL)
  4. Pulmonary edema
  5. Hypoglycemia (glucose in the blood <40mg/dL or clinic signs)
  6. Shock (PA systolic < 70 mm Hg in adults; < 50 in children)
  7. Spontaneous bleeding/Disseminated intravascular coagulation (CID)
  8. Recurrent generalized convulsions
  9. Acidemia/acidosis (clinic signs)
  10. Macroscopic hemoglobinuria
  11. Jaundice Laboratory tests for measuring some of these conditions may not be available at all study sites. If they are not, we will use clinical criteria of severe malaria at the discretion of the study physician
* Background of other chronic or severe diseases (e.g., heart, kidney, liver diseases, HIV/AIDS, severe malnutrition), determined clinically by medical history and physical examination
* Background of hypersensitivity to any of the drugs tested or used as an alternative treatment: AS, MQ, quinine or tetracycline/clindamycin
* Gestation (based on a serum pregnancy test or medical history) or desire to become pregnant during the study period, or not using any family planning method while being sexually active (confirmed by urine pregnancy test)
* Breastfeeding a child under 6 months old
* Have received antimalarial drugs in the previous 7 days
* Inability to eat or drink, vomiting (more than twice in the last 24 hours), recent history of seizures (one or more in the previous 24 hours), altered level of consciousness, inability to sit or stand
* Splenectomy background

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-06-18 (Actual); Primary Completion 2015-11-06 (Actual); Study Completion 2016-04-13 (Actual)

PRIMARY OUTCOMES:
Parasite clearance time | up to 72 hours after administration of artesunate
  Parasite clearance time assessed by microscopy and quantitative PCR

SECONDARY OUTCOMES:
Parasite reduction rates and ratios | 24, 48 hours after the first administration of artesunate
  Parasite reduction rates and ratios assessed by microscopy and quantitative PCR
Time for parasite count to fall | at least 24 hours
  Time for parasite count to fall to 50%, 90% and 99% of initial parasite density
Fever clearance time | at least 24 hours
  Time taken for temperature to fall below 37˚C and remain there for at least 24 hours
Gametocyte carriage rates | up to 14 days since the first administration of artesunate
  Gametocyte carriage rates assessed in person weeks up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Salomon Durand, Master, Principal Investigator — NAMRU 6
Locations (1):
- NAMRU 6, Iquitos, Loreto, Peru

REFERENCES:
- [Background] Durand S, Sihuincha M, Lachira A, Chaves J, Cabezas C. [A need to monitor P. falciparum resistance to artesunate in Peru]. Rev Peru Med Exp Salud Publica. 2012 Oct-Dec;29(4):579-80. doi: 10.1590/s1726-46342012000400028. No abstract available. Spanish. PMID 23338651
- [Background] de Oliveira AM, Chavez J, de Leon GP, Durand S, Arrospide N, Roberts J, Cabezas C, Marquino W. Efficacy and effectiveness of mefloquine and artesunate combination therapy for uncomplicated Plasmodium falciparum malaria in the Peruvian Amazon. Am J Trop Med Hyg. 2011 Sep;85(3):573-8. doi: 10.4269/ajtmh.2011.11-0250. PMID 21896825
- [Background] Gutman J, Green M, Durand S, Rojas OV, Ganguly B, Quezada WM, Utz GC, Slutsker L, Ruebush TK 2nd, Bacon DJ. Mefloquine pharmacokinetics and mefloquine-artesunate effectiveness in Peruvian patients with uncomplicated Plasmodium falciparum malaria. Malar J. 2009 Apr 9;8:58. doi: 10.1186/1475-2875-8-58. PMID 19358697
- [Background] Alker AP, Lim P, Sem R, Shah NK, Yi P, Bouth DM, Tsuyuoka R, Maguire JD, Fandeur T, Ariey F, Wongsrichanalai C, Meshnick SR. Pfmdr1 and in vivo resistance to artesunate-mefloquine in falciparum malaria on the Cambodian-Thai border. Am J Trop Med Hyg. 2007 Apr;76(4):641-7. PMID 17426163
- [Background] Wongsrichanalai C, Meshnick SR. Declining artesunate-mefloquine efficacy against falciparum malaria on the Cambodia-Thailand border. Emerg Infect Dis. 2008 May;14(5):716-9. doi: 10.3201/eid1405.071601. PMID 18439351